CLINICAL TRIAL: NCT00324038
Title: An Open, Randomised, Multicentre Study to Compare Buprenorphine Transdermal Delivery System (BTDS) With Standard Treatment in Elderly Subjects With OA of the Hip and/or Knee
Brief Title: Buprenorphine in the Treatment of Osteoarthritis (OA) in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Napp Pharmaceuticals Limited (Industry)
Responsible Party: Dr J Paul Schofield, Napp Pharmaceuticals Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-004279-39; BUP4004
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Results first posted 2010-03-30 (Estimated); Last update posted 2011-06-14 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
Keywords: OA; Elderly; Pain; OA of the hips and/or knees
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Buprenorphine; acetaminophen, codeine drug combination

ARMS (2):
- buprenorphine transdermal system (Experimental): Buprenorphine transdermal 7 day analgesic patch
  Interventions: Drug: Buprenorphine
- codeine paracetamol tablets (Active Comparator): codeine paracetamol combination tablets
  Interventions: Drug: Codeine paracetamol

INTERVENTIONS:
Drug: Buprenorphine — buprenorphine transdermal system 5, 10 and 20 mg
  Other Names: BuTrans/Norspan
  Arms: buprenorphine transdermal system
Drug: Codeine paracetamol — combination tablet of codeine and paracetamol taken orally 3 or 4 times daily. Dosage form ranges from 8/500, 15/500 and 30/500
  Other Names: Co-codamol tablets
  Arms: codeine paracetamol tablets

SUMMARY:
The primary objective is to compare buprenorphine transdermal delivery system (BTDS) with standard- treatment in subjects with osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* Either sex aged 65 or above
* Diagnosis of OA of the hip and/or knee
* Severe pain requiring step two medication
* Taking maximum dose of paracetamol

Exclusion Criteria:

* Painful disease of the joints other than OA
* Contraindication to buprenorphine, other opioids, patch adhesives or nonsteroidal anti-inflammatory agents (NSAIDS)
* Subjects taking cyclooxygenase (COX) II selective inhibitors

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 219 (Actual)
Dates: Start 2006-03; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof Philip Conaghan, Principal Investigator
Locations (1):
- Napp Pharmaceuticals Ltd, Cambridge, United Kingdom

REFERENCES:
- [Derived] Conaghan PG, O'Brien CM, Wilson M, Schofield JP. Transdermal buprenorphine plus oral paracetamol vs an oral codeine-paracetamol combination for osteoarthritis of hip and/or knee: a randomised trial. Osteoarthritis Cartilage. 2011 Aug;19(8):930-8. doi: 10.1016/j.joca.2011.03.011. Epub 2011 Apr 6. PMID 21477658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care. March 2006 to Aug 2007
Pre-assignment Details: Screening for patient eligibility
Groups:
- Buprenorphine Transdermal System: Buprenorphine transdermal system (patch)5mg, 10mg & 20mg worn for 7 days
- Co-codamol Tablets: combination tablet of codeine and paracetamol taken orally 3 or 4 times daily. Dosage form ranges from 8/500, 15/500 and 30/500
Period: Overall Study
Arm/Group | Buprenorphine Transdermal System | Co-codamol Tablets
Started | 110 | 109
Completed | 61 | 58
Not Completed | 49 | 51
Not completed — Adverse Event | 38 | 23
Not completed — Lack of Efficacy | 5 | 13
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine Transdermal System | Co-codamol Tablets | Total
Number analyzed (Participants) | 110 | 109 | 219
Age, Categorical [Count of Participants; unit: Participants] — Subjects over 60 years of age were recruited into the study. Initially study started with recruitment age of 65 but this was lowered by protocol amendment to 60 years of age.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 20 | 23 | 43
    >=65 years | 90 | 86 | 176
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 74 | 149
  Male | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Pain Scores - BS11 Pain Scores.
Description: The primary efficacy variable was the average daily pain score recorded on a Box Scale-11 pain scale in the evening. 0 = no pain and 10 = most pain imaginable. Subjects ticked the box from 0 - 10 which best describes their level of pain.
Time Frame: every day over a 12 week study duration.
Measure: Mean (Standard Deviation); unit: Box Scale 11 boxes
Arm/Group | Buprenorphine Transdermal System | Co-codamol Tablets
Number analyzed (Participants) | 61 | 58
Box Scale 11 boxes | 3 (1.31) | 3 (1.1)

ADVERSE EVENTS:
Description: Serious and non serious adverse events were collected/assessed but not serious adverse events
Arm/Group | Buprenorphine Transdermal System | Co-codamol Tablets
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No